CLINICAL TRIAL: NCT02670135
Title: Clinical Investigation of the Effects of Colgate Total Toothpaste as Compared to a Matching Placebo on Periodontal Disease and Systemic Inflammatory Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2014-09-CT-ISR-DB
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2015-06

CONDITIONS: Periodontal Disease; Systemic Inflammatory Markers
MeSH Terms: conditions — Periodontal Diseases | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triclosan free toothpaste (Placebo Comparator): Control toothpaste with no triclosan ingredients in a 1450 ppm sodium fluoride/silica base - matching placebo
  Interventions: Drug: Triclosan Free Toothpaste
- Triclosan containing toothpaste (Active Comparator): Active formula containing 0.3% triclosan in a1450 ppm sodium fluoride/silica base
  Interventions: Drug: Triclosan Containing Toothpaste

INTERVENTIONS:
Drug: Triclosan Containing Toothpaste — Active formula containing 0.3% triclosan in a1450 ppm sodium fluoride/silica base
  Other Names: Active comparator; Total Toothpaste
  Arms: Triclosan containing toothpaste
Drug: Triclosan Free Toothpaste — Control toothpaste with no triclosan ingredients in a 1450 ppm sodium fluoride/silica base - matching placebo
  Other Names: Control toothpaste
  Arms: triclosan free toothpaste

SUMMARY:
This is a single center, double blinded, randomized, controlled trial. Qualified subjects will be enrolled and randomized to either one of the two study groups: a) using 0.3% triclosan/copolymer/fluoride dentifrice twice daily - b) using a matching control dentifrice (copolymer/fluoride/no triclosan) twice daily.

DETAILED DESCRIPTION:
The objective of this study is to comparatively evaluate the effects of Colgate Total® toothpaste with triclosan (commercially sold in Israel) and triclosan-free matching placebo toothpaste on markers of inflammation in the bloodstream and to correlate these findings with periodontal disease status in the oral cavity, as determined by the parameters assessed. Periodontal parameters (periodontal pocket dept (PPD), Clinical Attachment loss (CAL)) will be assessed at baseline and after 2, 6 and 12 months of product use. Peripheral blood samples will be drawn from the subjects at baseline and after 2, 6 and 12 months to evaluate the effects of tooth brushing on systemic inflammatory markers (CRP, PGE2, IL-1β, TNF-α).

ELIGIBILITY:
Inclusion Criteria:

1. Subject males or females 18 to 50 years old.
2. Availability for the 12 months duration of the clinical research study.
3. Subject able and willing to follow study procedures and instructions.
4. Subject read, understood and signed an informed consent form.
5. Subject present with at least 20 natural teeth in the functional dentition (excluding third molars).
6. Initial probing pocket depth of >4mm in at least one tooth/quadrant.
7. Good general health.
8. Subjects willing to disclose information on medication.

Exclusion Criteria:

1. Subject with concomitant periodontal therapy 6 months prior to enrollment.
2. Subject with orthodontic appliances.
3. Subject chronically treated (i.e. two weeks or more) with any medication known to affect inflammation or periodontal status or within one month of the first examination*.
4. Subject treated with antibiotics within 3 months prior to enrollment.
5. Subject necessitating antibiotic prophylaxis.
6. Subject with active infectious diseases (hepatitis, human immunodeficiency virus or Tuberculosis) or subject is immunocompromised as determined by the Investigator*.
7. Subject with known allergy to oral care products or ingredients in oral care products.
8. Subject with gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque and calculus, or soft or hard tissue tumor of the oral cavity (determined by the examiner).
9. Subject diagnosed with aggressive periodontitis or acute necrotizing ulcerative gingivitis.
10. Participation in any other clinical study or test panel within the one month prior to entry into the study.
11. Subject pregnant at point of enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 303 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Periodontal Pocket Depth (PPD) | baseline
  PPD examination will be performed using a World Health Organization (WHO) Community Periodontal Index (CPI) periodontal probe in all teeth present as described by WHO (2013). The PPD examination is according to the pocket scores provided here: 0 = Absence of condition, 1 = Pocket 4-5mm, 2 = Pocket 6mm or more, 9 = Tooth excluded, X = Tooth not present (The lower the number the healthier the tissue)
Periodontal Pocket Depth (PPD) | 2 months
  PPD examination will be performed using a World Health Organization (WHO) Community Periodontal Index (CPI) periodontal probe in all teeth present as described by WHO (2013). The PPD examination is according to the pocket scores provided here: 0 = Absence of condition, 1 = Pocket 4-5mm, 2 = Pocket 6mm or more, 9 = Tooth excluded, X = Tooth not present (The lower the number the healthier the tissue)
Periodontal Pocket Depth (PPD) | 6 months
  PPD examination will be performed using a World Health Organization (WHO) Community Periodontal Index (CPI) periodontal probe in all teeth present as described by WHO (2013). The PPD examination is according to the pocket scores provided here: 0 = Absence of condition, 1 = Pocket 4-5mm, 2 = Pocket 6mm or more, 9 = Tooth excluded, X = Tooth not present (The lower the number the healthier the tissue)
Periodontal Pocket Depth (PPD) | 12 months
  PPD examination will be performed using a World Health Organization (WHO) Community Periodontal Index (CPI) periodontal probe in all teeth present as described by WHO (2013). The PPD examination is according to the pocket scores provided here: 0 = Absence of condition, 1 = Pocket 4-5mm, 2 = Pocket 6mm or more, 9 = Tooth excluded, X = Tooth not present (The lower the number the healthier the tissue)
Clinical Attachment Loss (CAL) | baseline
  Attachment lost will be measured from index teeth as described in WHO (2013). Loss of attachment is recorded by dividing the mouth in sextants, defined by tooth numbers: 18-14, 13-23, 24-28, 38-34, 33-43, and 44-48 Measurements will be recorded as: 0 = 0-3mm, 1 = 4-5mm (CEJ within black band), 2 = 6-8mm (CEJ between upper limit of black band and 8.5mm ring) 3 = 9-11mm (CEJ between 8.5mm ring and 11.5mm ring), 4 = 12mm and more (CEJ beyond 11.5mm ring), X = excluded, 9 = not recorded (The lower the number the healthier the tissue)
Clinical Attachment Loss (CAL) | 2 months
  Attachment lost will be measured from index teeth as described in WHO (2013). Loss of attachment is recorded by dividing the mouth in sextants, defined by tooth numbers: 18-14, 13-23, 24-28, 38-34, 33-43, and 44-48 Measurements will be recorded as: 0 = 0-3mm, 1 = 4-5mm (CEJ within black band), 2 = 6-8mm (CEJ between upper limit of black band and 8.5mm ring) 3 = 9-11mm (CEJ between 8.5mm ring and 11.5mm ring), 4 = 12mm and more (CEJ beyond 11.5mm ring), X = excluded, 9 = not recorded (The lower the number the healthier the tissue)
Clinical Attachment Loss (CAL) | 6 months
  Attachment lost will be measured from index teeth as described in WHO (2013). Loss of attachment is recorded by dividing the mouth in sextants, defined by tooth numbers: 18-14, 13-23, 24-28, 38-34, 33-43, and 44-48 Measurements will be recorded as: 0 = 0-3mm, 1 = 4-5mm (CEJ within black band), 2 = 6-8mm (CEJ between upper limit of black band and 8.5mm ring) 3 = 9-11mm (CEJ between 8.5mm ring and 11.5mm ring), 4 = 12mm and more (CEJ beyond 11.5mm ring), X = excluded, 9 = not recorded (The lower the number the healthier the tissue)
Clinical Attachment Loss (CAL) | 12 months
  Attachment lost will be measured from index teeth as described in WHO (2013). Loss of attachment is recorded by dividing the mouth in sextants, defined by tooth numbers: 18-14, 13-23, 24-28, 38-34, 33-43, and 44-48 Measurements will be recorded as: 0 = 0-3mm, 1 = 4-5mm (CEJ within black band), 2 = 6-8mm (CEJ between upper limit of black band and 8.5mm ring) 3 = 9-11mm (CEJ between 8.5mm ring and 11.5mm ring), 4 = 12mm and more (CEJ beyond 11.5mm ring), X = excluded, 9 = not recorded (The lower the number the healthier the tissue)
C Reactive Protein (CRP) | baseline
  C-reactive protein is a biomarker found in the blood and measures general levels of inflammation in your body. Inflammation plays a role in the initiation and progression of cardiovascular and potentially periodontal disease. The blood sample will be evaluated using Roche COBAS 6000 C501 system to quantify levels.
C Reactive Protein (CRP) | 2 months
  C-reactive protein is a biomarker found in the blood and measures general levels of inflammation in your body. Inflammation plays a role in the initiation and progression of cardiovascular and potentially periodontal disease. The blood sample will be evaluated using Roche COBAS 6000 C501 system to quantify levels.
C Reactive Protein (CRP) | 6 months
  C-reactive protein is a biomarker found in the blood and measures general levels of inflammation in your body. Inflammation plays a role in the initiation and progression of cardiovascular and potentially periodontal disease. The blood sample will be evaluated using Roche COBAS 6000 C501 system to quantify levels.
C Reactive Protein (CRP) | 12 months
  C-reactive protein is a biomarker found in the blood and measures general levels of inflammation in your body. Inflammation plays a role in the initiation and progression of cardiovascular and potentially periodontal disease. The blood sample will be evaluated using Roche COBAS 6000 C501 system to quantify levels.
Interleukin-1 Beta ( IL-1β) | baseline
  Inflammatory biomarker found in blood that may be a factor in oral tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer
Interleukin-1 Beta (IL-1β) | 2 months
  Inflammatory biomarker found in blood that may be a factor in oral tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer
Interleukin-1 Beta (IL-1β) | 6 months
  Inflammatory biomarker found in blood that may be a factor in oral tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer
Interleukin-1 Beta (IL- 1β) | 12 months
  Inflammatory biomarker found in blood that may be a factor in oral tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer
Tumor necrosis factor - alfa (TNF-α) | baseline
  TNF is a pro-inflammatory biomarker that is involved at an early stage inflammatory cascade and is released from mast cells in response to bacterial challenge. Drugs that block the action of TNF have been shown to be beneficial in reducing the inflammation in inflammatory diseases.
Tumor necrosis factor - alfa (TNF-α) | 2 months
  TNF is a pro-inflammatory biomarker that is involved at an early stage inflammatory cascade and is released from mast cells in response to bacterial challenge. Drugs that block the action of TNF have been shown to be beneficial in reducing the inflammation in inflammatory diseases.
Tumor necrosis factor - alfa (TNF-α) | 6 months
  TNF is a pro-inflammatory biomarker that is involved at an early stage inflammatory cascade and is released from mast cells in response to bacterial challenge. Drugs that block the action of TNF have been shown to be beneficial in reducing the inflammation in inflammatory diseases.
Tumor necrosis factor - alfa (TNF-α) | 12 months
  TNF is a pro-inflammatory biomarker that is involved at an early stage inflammatory cascade and is released from mast cells in response to bacterial challenge. Drugs that block the action of TNF have been shown to be beneficial in reducing the inflammation in inflammatory diseases.
Prostaglandin E2 (PGE 2) | baseline
  Inflammatory biomarker found in blood and may be a factor in tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer using Lithium-Heparin Plasma with an Indomethacin Inhibitor
Prostaglandin E2 (PGE 2) | 2 months
  Inflammatory biomarker found in blood and may be a factor in tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer using Lithium-Heparin Plasma with an Indomethacin Inhibitor
Prostaglandin E2 (PGE 2) | 6 months
  Inflammatory biomarker found in blood and may be a factor in tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer using Lithium-Heparin Plasma with an Indomethacin Inhibitor
Prostaglandin E2 (PGE 2) | 12 moths
  Inflammatory biomarker found in blood and may be a factor in tissue destruction as seen in periodontal disease. Levels will be quantified via the Automated Triturus ELISA Analyzer using Lithium-Heparin Plasma with an Indomethacin Inhibitor